CLINICAL TRIAL: NCT03532100
Title: Pivot-Flex Foot: Torsionally Adaptive Prosthesis for Individuals With Lower Limb Amputation
Brief Title: Pivot-Flex Foot: Optimal Coupling Ratio Between Transverse and Sagittal-plane Motions Using a Torsionally Adaptive Prosthesis for Individuals With Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: A2456-R; RX002456 Part 1 (Other: Department of Veterans Affairs, Rehabilitation R&D); I01RX002456-01A1 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Lower Extremity Amputation
Keywords: lower limb prosthesis; transtibial amputation; below knee amputation; biomechanics; gait

STUDY DESIGN:
Intervention Model Description: This within-subject, cross-over, factorial design study (3 arms x 5 intervention settings) aims to identify the optimal coupling ratio between transverse- and sagittal-plane motions using a torsionally adaptive prosthesis. The 3 arms including walking in a straight line (study visit 1) and walking in a circle with their lower limb prosthesis on the inside and outside of the circle (study visit 2). The order in which the participants walk around a circle with their prosthesis on the inside or the outside will be randomized. The study intervention, a torsionally adaptive prosthesis, can be set to 5 different settings (i.e., coupling ratios) including 0:0, 1:6, 1:4, 1:3, and 1:2 (transverse:sagittal). Within each arm, each participant will walk with the torsionally adaptive prosthesis set to the 5 different settings in random order. Participants will not be blinded to the arm but will be blinded to the intervention setting (coupling ratio).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Straight line walking (Experimental): All participants will walk in a straight line while wearing the study prosthesis.
  Interventions: Device: Torsionally adaptive prosthesis with 0:1 coupling ratio; Device: Torsionally adaptive prosthesis with 1:6 coupling ratio; Device: Torsionally adaptive prosthesis with 1:4 coupling ratio; Device: Torsionally adaptive prosthesis with 1:3 coupling ratio; Device: Torsionally adaptive prosthesis with 1:2 coupling ratio
- Circle walking with prosthesis inside (Experimental): All participants will walk around a 1-meter radius circle with their prosthesis on the inside of the circle.
  Interventions: Device: Torsionally adaptive prosthesis with 0:1 coupling ratio; Device: Torsionally adaptive prosthesis with 1:6 coupling ratio; Device: Torsionally adaptive prosthesis with 1:4 coupling ratio; Device: Torsionally adaptive prosthesis with 1:3 coupling ratio; Device: Torsionally adaptive prosthesis with 1:2 coupling ratio
- Circle walking with prosthesis outside (Experimental): All participants will walk around a 1-meter radius circle with their prosthesis on the outside of the circle.
  Interventions: Device: Torsionally adaptive prosthesis with 0:1 coupling ratio; Device: Torsionally adaptive prosthesis with 1:6 coupling ratio; Device: Torsionally adaptive prosthesis with 1:4 coupling ratio; Device: Torsionally adaptive prosthesis with 1:3 coupling ratio; Device: Torsionally adaptive prosthesis with 1:2 coupling ratio

INTERVENTIONS:
Device: Torsionally adaptive prosthesis with 0:1 coupling ratio — The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes. A coupling ratio (transverse:sagittal) of 0:1 means there will be no coupling between the transverse- and sagittal-plane motion. That is, regardless of any motion in the sagittal plane, there will be zero motion in the transverse plane.
Device: Torsionally adaptive prosthesis with 1:6 coupling ratio — The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes. A coupling ratio (transverse:sagittal) of 1:6 means there will be one degree of motion in the transverse plane for every six degrees of motion in the sagittal plane.
Device: Torsionally adaptive prosthesis with 1:4 coupling ratio — The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes. A coupling ratio (transverse:sagittal) of 1:4 means there will be one degree of motion in the transverse plane for every four degrees of motion in the sagittal plane.
Device: Torsionally adaptive prosthesis with 1:3 coupling ratio — The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes. A coupling ratio (transverse:sagittal) of 1:3 means there will be one degree of motion in the transverse plane for every three degrees of motion in the sagittal plane.
Device: Torsionally adaptive prosthesis with 1:2 coupling ratio — The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes. A coupling ratio (transverse:sagittal) of 1:2 means there will be one degree of motion in the transverse plane for every two degrees of motion in the sagittal plane.

SUMMARY:
When prescribing a prosthetic foot, clinicians face a dizzying array of choices as more than 200 different prosthetic feet are available. While these conventional prosthetic feet primarily function in the sagittal plane, the intact foot and ankle comprise a complex set of joints that allow rotation in multiple planes of motion. Some of these motions are coupled, meaning rotation in one plane induces motion in another. One such coupling is between the sagittal and transverse planes. For every step, plantar- and dorsi-flexion motion in the sagittal plane is coupled with external and internal rotation of the shank relative to the foot in the transverse plane. There is no prosthetic foot available for prescription that mimics this natural coupling.

To investigate the need for this coupling, the investigators have built a torsionally adaptive prosthesis where the coupling ratio between the transverse- and sagittal-planes can be independently controlled with a motor.

This research has one specific aim: to identify the optimal coupling ratio between transverse- and sagittal-plane motions using a novel, torsionally adaptive prosthesis for individuals with lower limb amputation. The investigators will conduct a human subject experiment wearing the motor-driven and computer controlled torsionally adaptive prosthesis. Individuals with lower limb amputation will be asked to walk in a straight line and in both directions around a circle while the coupling ratio between transverse- and sagittal-plane motions is varied between trials. Participants will be blinded to the coupling ratio.

The investigators hypothesize that: (1) a coupling ratio exists that minimizes undesirable transverse-plane socket torque and (2) there will be a coupling ratio that individuals with lower limb amputation prefer.

DETAILED DESCRIPTION:
The human ankle is a complex mechanism that does not behave like a simple hinge. Instead, rotations in all three axes are allowed and some are coupled together. In particular, the axis of rotation of the talo-crural joint during ankle flexion is inclined downwards and laterally relative to horizontal, and the rotation ranges from 10 to 26 degrees among individuals. This rotation couples plantar- and dorsi-flexion motion with external and internal rotation of the shank relative to the foot, respectively. This feature of the natural limb has not been replicated in prosthetic feet and ankles.

Lower limb amputees take thousands of steps on their prosthesis each day and none feature coupled motion between the transverse- and sagittal-planes. The absence of this natural coupling may be related to the high incidence of residual limb soft tissue injuries, the need for compensatory gait, and overall dissatisfaction with their prostheses.

Transverse rotation adapters, consisting of simple torsional springs, are available for prescription. These devices can increase transverse-plane rotations and decrease transverse-plane torques, but their use is not widespread and if excessively compliant, may reduce gait stability. Cost, weight, prosthesis build height, and the inability for the user to adjust the stiffness may all play a role in their lack of adoption, but it may also be that the transverse-plane rotation is not coupled with the sagittal-plane. With these devices, motion only occurs in the transverse-plane when a transverse-plane torque is applied.

This research has one specific aim: to identify the optimal coupling ratio between transverse- and sagittal-plane motions using a novel, torsionally adaptive prosthesis for individuals with lower limb amputation. The investigators will fit a sample population of unilateral transtibial amputees with the motor-driven and computer controlled torsionally adaptive prosthesis.

Participants perform three activities: walking in a straight line (study visit 1) and in both directions around a circle (study visit 2). During each of these three activities, the torsionally adaptive prosthesis will be set to five different coupling ratios in random order. Participants will be blinded to the coupling ratio.

The general hypotheses for this study are: (H1) a coupling ratio exists between 0 (no coupling) to 1:2 (one degree of transverse-plane motion for every two degrees of sagittal-plane motion) that minimizes transverse-plane socket torque and (H2) an amputee preferred coupling ratio will exist within this range.

This research will discover how best to couple transverse- and sagittal-plane motion in the prostheses of lower limb amputees.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* Been fit with a prosthesis and used it for at least six months
* Wear the prosthesis for four or more hours on an average day
* Prescribed prosthesis can accommodate fitment of the study prosthetic components to be tested (determined at initial visit)

Exclusion Criteria:

* Improper fit and suspension with current prosthesis and one cannot be achieved with clinical resources (determined at initial visit)
* Current skin irritation or injury on residual limb
* Osteoarthritis, injury, or pain that interferes with walking ability
* Currently incarcerated
* Pregnant (determined via self-report)
* Inadequate cognitive function or language proficiency to consent to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset in machine-readable format will be created and shared for all individual participant data (IPD) that underlie results in a publication. The investigators will follow 164.514(a) of the HIPAA Privacy Rule for de-identification of IPD.
Time Frame: Within six months after publication of final study findings.
Access Criteria: Open access through PubMed Central, SimTK, PhysioNet, or other similar open-source data repository websites. The investigators will work with manuscript publishers when possible to link the final study data sets to an appendix of supplemental materials on the publisher websites.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two enrolled participants decided they were no longer interested in participating before beginning the study protocol. One enrolled participant had a long residual limb and could not accommodate the build height of the study intervention.
Groups:
- Individuals With a Lower Limb Prosthesis: In this cross-over study, all subjects were asked to perform 3 activities:
  1. Walking in a straight line while wearing the study intervention (prosthesis),
  2. Walking around a 2-meter diameter circle with the study intervention (prosthesis) on the inside of the circle, and
  3. Walking around a 2-meter diameter circle with the study intervention (prosthesis) on the outside of the circle.
  While performing each of these activities, the study intervention was set to 5 different settings (5 sagittal:transverse coupling ratio, 1:0, 6:1, 4:1, 3:1, and 2:1). These settings were block randomized and blinded to the participant.
  The study was conducted over two visits with overnight rest in between each visit. During the first study visit, participants performed the walking in a straight line activity. During the second study visit, participants walked around a 2-meter diameter circle with the study intervention (prosthesis) on the inside and the outside of the circle. The order in which the participants walked with the study intervention (prosthesis) on the inside or the outside of the circle was randomized.
Period: Overall Study
Arm/Group | Individuals With a Lower Limb Prosthesis
Started | 11
** Straight Line Walking | 11
Straight Line Walking With 0:1 Coupling Ratio | 11
Straight Line Walking With 1:6 Coupling Ratio | 11
Straight Line Walking With 1:4 Coupling Ratio | 11
Straight Line Walking With 1:3 Coupling Ratio | 11
Straight Line Walking With 1:2 Coupling Ratio | 11
** Circle Walking With Prosthesis on the Inside | 11
Circle Walking With Prosthesis on the Inside and 0:1 Coupling Ratio | 11
Circle Walking With Prosthesis on the Inside and 1:6 Coupling Ratio | 11
Circle Walking With Prosthesis on the Inside and 1:4 Coupling Ratio | 11
Circle Walking With Prosthesis on the Inside and 1:3 Coupling Ratio | 11
Circle Walking With Prosthesis on the Inside and 1:2 Coupling Ratio | 11
** Circle Walking With Prosthesis on the Outside | 10 (An intervention malfunction prevented one subject from performing the walk around a 2-meter diameter circle with the prosthesis on the outside.)
Circle Walking With Prosthesis on the Outside and 0:1 Coupling Ratio | 10
Circle Walking With Prosthesis on the Outside and 1:6 Coupling Ratio | 10
Circle Walking With Prosthesis on the Outside and 1:4 Coupling Ratio | 10
Circle Walking With Prosthesis on the Outside and 1:3 Coupling Ratio | 10
Circle Walking With Prosthesis on the Outside and 1:2 Coupling Ratio | 10
Completed | 10
Not Completed | 1
Not completed — Intervention malfunction | 1

BASELINE CHARACTERISTICS:
Groups:
- Individuals With a Lower Limb Amputation: All participants were block randomized to the order in which they walked in a straight line, walked around a 2m diameter circle with their prosthesis on the inside of the circle, and walked around a 2m diameter circle with their prosthesis on the outside of the circle. Additionally, the order of the sagittal:transverse coupling ratio of 1:0, 6:1, 4:1, 3:1, and 2:1 were also block randomized and blinded to the participant.
Arm/Group | Individuals With a Lower Limb Amputation
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Transverse-plane Prosthetic Socket Torque Normalized to Body Mass
Description: Peak transverse-plane prosthetic socket torque measured while walking normalized to body mass
Time Frame: During walking trials for each coupling ratio
Measure: Mean (Standard Error); unit: Nm/kg
Groups:
- Straight Line Walking: All participants will walk in a straight line while wearing the study prosthesis. The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes.
  Torsionally adaptive prosthesis with 0:1 coupling ratio. A coupling ratio (transverse:sagittal) of 0:1 means there will be no coupling between the transverse- and sagittal-plane motion. That is, regardless of any motion in the sagittal plane, there will be zero motion in the transverse plane.
  Torsionally adaptive prosthesis with 1:6 coupling ratio. A coupling ratio (transverse:sagittal) of 1:6 means there will be one degree of motion in the transverse plane for every six degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:4 coupling ratio. A coupling ratio (transverse:sagittal) of 1:4 means there will be one degree of motion in the transverse plane for every four degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:3 coupling ratio. A coupling ratio (transverse:sagittal) of 1:3 means there will be one degree of motion in the transverse plane for every three degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:2 coupling ratio. A coupling ratio (transverse:sagittal) of 1:2 means there will be one degree of motion in the transverse plane for every two degrees of motion in the sagittal plane.
- Circle Walking With Prosthesis Inside: All participants will walk around a 1-meter radius circle with their prosthesis on the inside of the circle. The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes.
  Torsionally adaptive prosthesis with 0:1 coupling ratio. A coupling ratio (transverse:sagittal) of 0:1 means there will be no coupling between the transverse- and sagittal-plane motion. That is, regardless of any motion in the sagittal plane, there will be zero motion in the transverse plane.
  Torsionally adaptive prosthesis with 1:6 coupling ratio. A coupling ratio (transverse:sagittal) of 1:6 means there will be one degree of motion in the transverse plane for every six degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:4 coupling ratio. A coupling ratio (transverse:sagittal) of 1:4 means there will be one degree of motion in the transverse plane for every four degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:3 coupling ratio. A coupling ratio (transverse:sagittal) of 1:3 means there will be one degree of motion in the transverse plane for every three degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:2 coupling ratio. A coupling ratio (transverse:sagittal) of 1:2 means there will be one degree of motion in the transverse plane for every two degrees of motion in the sagittal plane.
- Circle Walking With Prosthesis Outside: All participants will walk around a 1-meter radius circle with their prosthesis on the outside of the circle. The torsionally adaptive prosthesis can be programmed to couple the motion between the transverse- and sagittal-planes.
  Torsionally adaptive prosthesis with 0:1 coupling ratio. A coupling ratio (transverse:sagittal) of 0:1 means there will be no coupling between the transverse- and sagittal-plane motion. That is, regardless of any motion in the sagittal plane, there will be zero motion in the transverse plane.
  Torsionally adaptive prosthesis with 1:6 coupling ratio. A coupling ratio (transverse:sagittal) of 1:6 means there will be one degree of motion in the transverse plane for every six degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:4 coupling ratio. A coupling ratio (transverse:sagittal) of 1:4 means there will be one degree of motion in the transverse plane for every four degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:3 coupling ratio. A coupling ratio (transverse:sagittal) of 1:3 means there will be one degree of motion in the transverse plane for every three degrees of motion in the sagittal plane.
  Torsionally adaptive prosthesis with 1:2 coupling ratio. A coupling ratio (transverse:sagittal) of 1:2 means there will be one degree of motion in the transverse plane for every two degrees of motion in the sagittal plane.
Arm/Group | Straight Line Walking | Circle Walking With Prosthesis Inside | Circle Walking With Prosthesis Outside
Number analyzed (Participants) | 11 | 11 | 10
Nm/kg
  Sagittal:transverse coupling ratio 1:0 | 0.299 (0.025) | 0.340 (0.026) | 0.306 (0.026)
  Sagittal:transverse coupling ratio 6:1 | 0.292 (0.013) | 0.324 (0.023) | 0.306 (0.026)
  Sagittal:transverse coupling ratio 4:1 | 0.312 (0.011) | 0.331 (0.023) | 0.322 (0.025)
  Sagittal:transverse coupling ratio 3:1 | 0.323 (0.012) | 0.343 (0.019) | 0.336 (0.021)
  Sagittal:transverse coupling ratio 2:1 | 0.350 (0.019) | 0.349 (0.021) | 0.358 (0.021)
Statistical Analysis 1: Comparison: Straight Line Walking; Hypothesis testing for the association between outcome and coupling ratio was carried out using conditional F-tests with degrees of freedom estimated using the Kenward-Roger method; Test type: Superiority; p = 0.029, Regression, Linear
Statistical Analysis 2: Comparison: Straight Line Walking; 6:1 versus 3:1; Test type: Superiority; p = 0.047, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method
Statistical Analysis 3: Comparison: Straight Line Walking; 6:1 versus 2:1; Test type: Superiority; p = 0.016, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method
Statistical Analysis 4: Comparison: Circle Walking With Prosthesis Inside; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.340, Regression, Linear
Statistical Analysis 5: Comparison: Circle Walking With Prosthesis Outside; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, Regression, Linear
Statistical Analysis 6: Comparison: Circle Walking With Prosthesis Outside; 6:1 versus 3:1; Test type: Superiority; p = 0.036, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method
Statistical Analysis 7: Comparison: Circle Walking With Prosthesis Outside; 6:1 versus 2:1; Test type: Superiority; p = 0.028, Regression, Linear — Pairwise hypothesis testing was carried out with adjustments for multiple comparisons using Tukey's method

2. Secondary Outcome: Satisfaction With the Prosthesis
Description: An 11-point Likert scale will be used to record the subject's perception of satisfaction with the prosthesis after completing the trials for each coupling ratio. Participants will be asked to rate their satisfaction with the prosthesis on a 0 - 10 scale. Zero represented the most uncomfortable socket fit the subject could imagine, and ten represented the most comfortable socket fit.
Time Frame: Immediately following walking trials for each coupling ratio
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Straight Line Walking | Circle Walking With Prosthesis Inside | Circle Walking With Prosthesis Outside
Number analyzed (Participants) | 11 | 11 | 10
score on a scale
  Sagittal:transverse coupling ratio 1:0 | 8.0 (1.3) | 7.5 (1.3) | 7.7 (1.7)
  Sagittal:transverse coupling ratio 6:1 | 8.2 (1.3) | 7.9 (1.1) | 7.9 (1.2)
  Sagittal:transverse coupling ratio 4:1 | 8.0 (1.0) | 7.1 (1.7) | 7.4 (1.3)
  Sagittal:transverse coupling ratio 3:1 | 7.7 (1.2) | 7.5 (0.7) | 7.8 (1.1)
  Sagittal:transverse coupling ratio 2:1 | 8.5 (1.0) | 8.1 (1.3) | 7.7 (1.5)

ADVERSE EVENTS:
Time Frame: 1 week
Description: In this study, subjects only wore the study intervention while in the laboratory under supervision of laboratory staff. Because the 3 arms (activities) and the 5 intervention settings could be quickly changed, adverse events for all arms and interventions were combined.
Groups:
- Individuals With a Lower Limb Amputation: All participants performed walking in a straight line (study visit 1) and walking in a circle with their lower limb prosthesis on the inside and outside of the circle (study visit 2). The order in which the participants walked around a circle with their prosthesis on the inside or the outside was randomized. During each walking activity, the participants experienced each of the five different intervention settings (i.e., coupling ratios) in random order. Participants were blinded to the intervention setting.
Arm/Group | Individuals With a Lower Limb Amputation
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03532100/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT03532100/SAP_001.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT03532100/ICF_002.pdf